CLINICAL TRIAL: NCT01794468
Title: A New Monitor to Measure Dermal Blood Flow in Critically Ill Patients: a Preliminary Study
Acronym: MDBF-CIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Pierre singer, Professor , MD, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3030
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Positive-Pressure Respiration, Intrinsic; Critically Ill Patients
Keywords: Dermal blood flow; critically ill
MeSH Terms: conditions — Positive-Pressure Respiration, Intrinsic; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study group-Dermal blood flow measurements (Experimental): Dermal blood flow was measured with the Dermal Blood Flow (DBF) monitor
  Interventions: Other: Dermal blood flow measurements

INTERVENTIONS:
Other: Dermal blood flow measurements — Dermal blood flow was measured with the Dermal Blood Flow (DBF) monitor (I.S. MedTech, Israel), which consists of a skin probe and a measuring and control feedback unit.

SUMMARY:
Background: Conditions of reduced perfusion are characterized by redistribution of blood flow away from the skin to more vital organs.

Study Objectives: To assess the efficacy of a non-invasive, dermal blood flow (DBF) monitor in detecting changes in perfusion in critically ill patients.

Preliminary Study

Study Population: critically ill patients in a general ICU

DETAILED DESCRIPTION:
DBF, finger plethysmography and invasive mean arterial pressure (MAP) were recorded over an 8-hour period. DBF was measured using the I.S. MedTech DBF monitor, based on the hot-wire principle of thermal balance of a heater cooled by a moving medium, via a skin probe placed on the anterior chest wall. Sensitivity was evaluated by visual inspection during active states, either induced, e.g. fluid administration, or spontaneous, e.g. altered hemodynamics. Specificity was evaluated during stable states (minimal fluctuations of MAP and no active interventions applied or required). Data are expressed in terms of standard deviation (SD) and of the difference (SDD) between the MAP and each of the tested methods.

ELIGIBILITY:
Inclusion Criteria:

* All patients were ventilated and sedated during an 8-hour period of measurement

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-06; Primary Completion 2005-04 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Dermal blood flow measurements | over an 8-hour period
  DBF monitor - non-invasive method for detecting changes in perfusion in critically ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cohen, Professor,MD, Study Chair — ICU dep't, Rabin MC,Petah Tikva, Israel; Pierre Singer, Professor,MD, Principal Investigator — ICU dep't, Rabin MC,Petah Tikva, Israel
Locations (1):
- ICU dep't , Rabin MC, Petah Tikva, Israel